CLINICAL TRIAL: NCT06369922
Title: Transcutaneous Electrical Nerve Stimulation Analgesia During Outpatient Urethral Bulking for Stress Urinary Incontinence.
Brief Title: TENS Analgesia During Outpatient Urethral Bulking for Stress Urinary Incontinence.
Acronym: TENSUB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jared Matthew Floch, Fellow, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00009315
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Stress Incontinence Female; Urinary Incontinence; Urinary Incontinence,Stress; Pain; Pain Acute
Keywords: TENS; pain; Transcutaneous Electrical Nerve Stimulation Analgesia
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Pain; Acute Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TENS (Experimental): In the active treatment group, the TENS unit will remain on up to 30 minutes (10 minutes pre-procedure, during the procedure and during the questionnaires).
  Interventions: Procedure: TENS
- Control TENS (Sham Comparator): The sham stimulation group will undergo the same procedure; however, the TENS stimulation current will be reduced to a minimal detectable level and turned off after 20 seconds.
  Interventions: Procedure: Control TENS

INTERVENTIONS:
Procedure: TENS — This device will then be used for deep transcutaneous nerve stimulation at the T10-L1 and S2-S4 levels. The device will be placed and activated 5 minutes before the procedure. and the device will remain active during the procedure and will be turned off as soon as the procedure is complete (the procedure typically takes 5-15 minutes). The TENS units have pre-program settings, improving convenience, reproducibility, and reliability. Study staff will be instructed to perform TENS using an "Acupuncture" mode on the provided TENS units. The amplitude will be adjusted to a comfortable sensation that does not cause pain using adhesive electrodes. One TENS unit is able to support 4 TENS electrodes. The TENS electrodes (8 cm x 5 cm) will be placed on bilateral paraspinal muscles. The intensity of the stimulation (Hz) will be adjusted to the subjective comfort of the subject.
  Arms: Active TENS
Procedure: Control TENS — This device will then be used for deep transcutaneous nerve stimulation at the T10-L1 and S2-S4 levels. The device will be placed and activated 5 minutes before the procedure. and the device will remain active during the procedure and will be turned off as soon as the procedure is complete (the procedure typically takes 5-15 minutes). The TENS units have pre-program settings, improving convenience, reproducibility, and reliability. Study staff will be instructed to perform TENS using an "Acupuncture" mode on the provided TENS units. The amplitude will be adjusted to a comfortable sensation that does not cause pain using adhesive electrodes. One TENS unit is able to support 4 TENS electrodes. The TENS electrodes (8 cm x 5 cm) will be placed on bilateral paraspinal muscles. The intensity of the stimulation (Hz) will be adjusted to the subjective comfort of the subject.
  Arms: Control TENS

SUMMARY:
This will be a double-blind randomized control trial in women with stress urinary incontinence who are undergoing an outpatient transurethral bulking procedure for stress urinary incontinence. Subjects will be identified by the University of Rochester urologists and urogynecologists participating in the study who currently oversee stress incontinence care. Subjects will be randomized into two groups. One group will be undergoing the cystoscopy with transcutaneous electrical nerve stimulation (TENS) for analgesia, and the second group will have the cystoscopy with placebo TENS.

DETAILED DESCRIPTION:
This will be a double-blind randomized control trial in women with stress urinary incontinence who are undergoing outpatient transurethral bulking procedures. These subjects will be identified by the University of Rochester urologists and urogynecologists participating in the study, who oversee the patient's stress urinary incontinence management. The subjects will be asked to participate in this research project when the doctor is offering options for their SUI treatment.

Subjects will be randomized into two groups. One group will undergo transurethral bulking with TENS for analgesia, and the second group will have the procedure performed with placebo TENS. The application of the TENS device will be performed by a study team member who will know to what group the patient was randomized. Both groups will be given the VAS, satisfaction scale, and 5-point Likert scale questionnaires to be answered before, during, and after they undergo treatment on the scheduled day of the procedure.

The primary outcome will be a change in the VAS pain measurement. Investigators hypothesized that TENS used during transurethral bulking injections would result in a 10-mm decrease in VAS compared to placebo TENS.

Secondary outcomes will be:

1. A discrete 5-point Likert Scale to assess the internal consistency of the pain rating within the study
2. A satisfaction 10-point scale questionnaire
3. Rate of side effects to the use of TENS (skin irritation, pain or burning at electrode site) and transurethral bulking injections (vasovagal symptoms: dizziness, nausea, vomiting, shoulder pain, vertigo, sweating, fainting),
4. Length of procedure.

ELIGIBILITY:
Inclusion Criteria:

* • Women, Age ≥18 years

  * Diagnosis of SUI
  * Scheduled to undergo transurethral bulking in the office
  * Able to read/write English

Exclusion Criteria:

* • Cutaneous damage such as ulcers or broken skin on target treatment area

  * Currently implanted cardiac pacemaker or defibrillator
  * Pre-procedural use of opioids for pain management, less than 8 hours from last dose
  * Participants with altered sensation below the umbilicus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean pain measured by Visual Analog Scale (VAS) | Before procedure
  The VAS for pain consists of a 100-mm-long horizontal line where 0-mm equals no pain and 100-mm equals worst possible pain.
Mean pain measured by Visual Analog Scale (VAS) | Approximately 2-5 minutes into the procedure
  The VAS for pain consists of a 100-mm-long horizontal line where 0-mm equals no pain and 100-mm equals worst possible pain.
Mean pain measured by Visual Analog Scale (VAS) | within 10 minutes after procedure
  The VAS for pain consists of a 100-mm-long horizontal line where 0-mm equals no pain and 100-mm equals worst possible pain.

SECONDARY OUTCOMES:
Mean pain measured by Likert scale | before procedure
  A discrete, 5-point verbal Likert scale including the following options: "no pain", "minimal pain", "moderate pain", "severe pain" and "worst pain possible" will be asked to patients
Mean pain measured by Likert scale | Approximately 2-5 minutes into the procedure
  A discrete, 5-point verbal Likert scale including the following options: "no pain", "minimal pain", "moderate pain", "severe pain" and "worst pain possible" will be asked to patients
Mean pain measured by Likert scale | within 10 minutes after procedure
  A discrete, 5-point verbal Likert scale including the following options: "no pain", "minimal pain", "moderate pain", "severe pain" and "worst pain possible" will be asked to patients
Number of participants with side effects | within 10 minutes after procedure
  A check list of vasovagal symptoms will be handed to the study team member to complete if the subject reports any light headedness, nausea or sweating.
Mean satisfaction with the procedure | within 10 minutes after procedure
  A 1-10 point satisfaction scale will be used where 10 indicates higher satisfaction.
TENS or NO TENS | within 10 minutes after procedure
  Number of participants who guessed correctly whether they were given the active TENS or placebo TENS

CONTACTS AND LOCATIONS:
Locations (1):
- Pelvic Health and Continence Specialties, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided